CLINICAL TRIAL: NCT02336217
Title: Glycemic Emergency Management (GEM); An App for Rapid Response to Hypoglycemic and Hyperglycemic Situations
Acronym: GEMApp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Henry Driscoll, MD, Chief, section of Endocrinology, Marshall University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 574049
Record Dates: First submitted 2014-11-14; First posted 2015-01-12 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Functioning App (Experimental): These subjects have the complete algorithm functioning and communicated via the App.
  Interventions: Other: Experimental Group instructions for glucose management via App
- Non-functioning App (Placebo Comparator): These subjects receive routine instructions via the App but not the complete algorithm.
  Interventions: Other: Placebo Comparator general instructions

INTERVENTIONS:
Other: Experimental Group instructions for glucose management via App — The Experimental Group receives individually calculated instructions for glucose management management via the App.
  Arms: Functioning App
Other: Placebo Comparator general instructions — The Placebo Comparator Group receives general instructions but not the complete management algorithm
  Arms: Non-functioning App

SUMMARY:
The purpose of this pilot study is to determine the utility of an algorithm for better glucose control in diabetic patients communicated via an App to help improve outcomes and reduce urgent care and ER visits as well as improve A1C and quality of life.

DETAILED DESCRIPTION:
The aim of the study is to determine the impact of GEM (glycemic emergency management device-app) in reducing the frequency and severity of hypoglycemia episodes in persons with diabetes. Other objectives include: to determine whether the GEM system leads to improved glucose control (as measured by HbA1c) during participation in the pilot, to determine whether the GEM can be used as a cost effective solution in reducing ER and urgent care visits, to determine the difference in ADDQOL scores between persons with a functioning GEM system and those with a placebo device. The Study hypothesis is as follows: There wil be significant differences in number of hypoglycemic events, ER and urgent care visits, A1C, as well as quality of life as measured by the ADDQOL scores between persons with diabetes who have the functioning GEM device in their smart phones and those that do not have such a device installed in their smart phones.

The purpose of this pilot study is to determine the utility of this application to help improve outcomes and reduce urgent care and ER visits as well as improve A1C and quality of life in persons with diabetes. This approach may be a paradigm shift in the rapidly detecting, monitoring, intervening and managing the acute diabetic complications of hypoglycemia, hyperglycemia and diabetic ketoacidosis. Spiraling health care costs are a major concern to the economy of the US. New measures have been introduced in the Affordable Care Act to improve the efficiency of the health care delivery system. There is more emphasis on preventive health care services. Our study is a step in that direction since it utilizes existing smart phone technology and converts it into a medical device which can be of invaluable help to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes on therapeutic treatment other than just lifestyle changes
* Treatment by Marshall Internal Medicine Department
* Have a smart phone
* At least 6th grade education level

Exclusion Criteria:

* Pregnant women
* Cognitive impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of hypoglycemic episodes | 6 months

SECONDARY OUTCOMES:
A1c level | 6 months
Number of Emergency Room, Urgent Care, or Walk-In Clinic visits | 6 months
ADDQOL score | 6 months
  Quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall Health, Huntington, West Virginia, United States